CLINICAL TRIAL: NCT01955967
Title: The Effect of Intravenous Lidocaine on Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Relief & Palliative Care Center, Athens, Greece (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Trigeminal Neuralgia
Keywords: Effect; Lidocaine
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Lidocaine (Other)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
The aim of this randomized double blind, placebo controlled, crossover study is to investigate in a prospective way the effect of lidocaine in patients with trigeminal neuralgia. Included patients will undergo four weekly sessions, two of which with lidocaine (5mgs/kg) and two with placebo infusions administered over 60 minutes. Effect will be measured with pain diaries and visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

(1) confirmed diagnosis of TN according to IASP definition, (2) age equal to or greater than 18 years, (3) visual analogue scale (VAS) score equal to or greater than 3 (out of a maximum 10), (4) DN4 score equal to or greater than 4 (out of a maximum 10), (5) having received the recommended medications for TN (antiepileptics, spasmolytics, opioids, anti-inflammatory and simple analgesic drugs) for an adequate period without therapeutic results, (6) TN duration of at least 12 months, (8) no history of allergy to lidocaine, (9) no history of substance abuse, (10) absence of severe psychiatric diseases, (11) not being pregnant, (12) not lactating, (13) absence of severe cardiac, hepatic and renal decease, and (14) be willing to provide a written informed consent to undergo the experimental procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24h

REFERENCES:
- [Derived] Stavropoulou E, Argyra E, Zis P, Vadalouca A, Siafaka I. The Effect of Intravenous Lidocaine on Trigeminal Neuralgia: A Randomized Double Blind Placebo Controlled Trial. ISRN Pain. 2014 Mar 10;2014:853826. doi: 10.1155/2014/853826. eCollection 2014. PMID 27335883